CLINICAL TRIAL: NCT03098641
Title: Transvaginal Treatment of Anterior and Apical Genital Prolapses Using an Ultra Lightweight Mesh: Restorelle® Direct FixTM: a Retrospective Study on Feasibility and Morbidity.
Brief Title: Smartmesh Technology in Pelvic Floor Repair Procedures
Acronym: Restorelle
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016/P05/179
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2019-06-03 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pelvic organ prolapse repair — Surgery to repair pelvic organ prolapse through the vagina using stitches with the addition of surgical mesh.

SUMMARY:
Pelvic organ prolapse repair involves conservative treatments and surgical treatments. Conservative treatments are for patients with moderate prolapse. Treatment of symptomatic prolapse remains essentially surgical. According to detailed medical history and a thorough physical exam, surgical techniques may be performed by high abdominal, low vaginal or mixed routes with or without the use of a reinforcing implant. Restorelle Direct Fix is indicated for transvaginal anterior and posterior surgical repair either as mechanical support or as reinforcement of pelvic floor defects. Advantages and disadvantages of vaginal prostheses are known but only limited data have been reported on the use of Restorelle® in the treatment of pelvic organ prolapse. This study is designed to collect data on the safety and efficacy of Restorelle® Direct Fix in pelvic organ prolapse repair.

DETAILED DESCRIPTION:
Between January 2013 and December 2016, in the participating centers, all adult women who underwent surgery to repair pelvic organ prolapse (recurrent or not) through the vagina with the addition of anterior and/or posterior Restorelle Direct Fix prosthesis are eligible. Collected data are about the peri-operative period and the data available at the last consultation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* woman who underwent surgery to repair pelvic organ prolapse (recurrent or not) through the vagina with the addition of anterior and/or posterior Restorelle Direct Fix prosthesis
* informed and not opposed to the use of her data

Exclusion Criteria:

* Opposed to the use of her data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women who underwent surgery to repair pelvic organ prolapse (recurrent or not) through the vagina with the addition of anterior and/or posterior Restorelle Direct Fix prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ferry, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (16):
- France (16):
  - CH Dunkerque, Grande-Synthe
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - Clinique Saint Ame, Lambres-lez-Douai
  - CH de Laon, Laon
  - Clinique Jules Verne, Nantes
  - CHU Nîmes, Nîmes
  - Hôpital des Diaconesses, Paris
  - Hôpital Kremlin-Bicêtre, Paris
  - CH de Cornouaille, Quimper
  - Clinique St Michel et St Anne, Quimper
  - Polyclinique de Courlancy, Reims
  - Clinique la Sagesse, Rennes
  - CH Robert Pax, Sarreguemines
  - Agyl, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpitaux du Léman, Thonon-les-Bains

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Le Normand L, Cosson M, Cour F, Deffieux X, Donon L, Ferry P, Fatton B, Hermieu JF, Marret H, Meurette G, Cortesse A, Wagner L, Fritel X. [Clinical practice guidelines: Summary of recommendations for first surgical treatment of female pelvic organ prolapse by 5 French academic societies: AFU, CNGOF, SIFUD-PP, SNFCP, and SCGP]. Prog Urol. 2016 Jul;26 Suppl 1:S1-7. doi: 10.1016/S1166-7087(16)30424-9. French. PMID 27595623
- [Background] Khunda A, Vashisht A, Cutner A. New procedures for uterine prolapse. Best Pract Res Clin Obstet Gynaecol. 2013 Jun;27(3):363-79. doi: 10.1016/j.bpobgyn.2012.12.004. Epub 2013 Jan 5. PMID 23298608
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] Persu C, Chapple CR, Cauni V, Gutue S, Geavlete P. Pelvic Organ Prolapse Quantification System (POP-Q) - a new era in pelvic prolapse staging. J Med Life. 2011 Jan-Mar;4(1):75-81. Epub 2011 Feb 25. PMID 21505577
- [Background] Lousquy R, Costa P, Delmas V, Haab F. [Update on the epidemiology of genital prolapse]. Prog Urol. 2009 Dec;19(13):907-15. doi: 10.1016/j.purol.2009.09.011. Epub 2009 Nov 4. French. PMID 19969258
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Marjoribanks J. Transvaginal mesh or grafts compared with native tissue repair for vaginal prolapse. Cochrane Database Syst Rev. 2016 Feb 9;2(2):CD012079. doi: 10.1002/14651858.CD012079. PMID 26858090
- [Result] Ferry P, Bertherat P, Gauthier A, Villet R, Del Piano F, Hamid D, Fernandez H, Broux PL, Salet-Lizee D, Vincens E, Ntshaykolo P, Debodinance P, Pocholle P, Thirouard Y, de Tayrac R. Transvaginal treatment of anterior and apical genital prolapses using an Ultra lightweight mesh: Restorelle(R) Direct Fix. A retrospective study on feasibility and morbidity. J Gynecol Obstet Hum Reprod. 2018 Nov;47(9):443-449. doi: 10.1016/j.jogoh.2018.06.001. Epub 2018 Jun 18. PMID 29920380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2013 and December 2016, in 10 secondary and tertiary French care centres
Pre-assignment Details: Patients were excluded if they did not attend their follow up visit within 30 days of surgery.
Groups:
- Pelvic Organ Prolapse Repair: Adult women who had vaginal repair of pelvic organ prolapse (recurrent or not) planned with anterior Restorelle® Direct FixTM mesh (with or without posterior mesh)
Period: Overall Study
Arm/Group | Pelvic Organ Prolapse Repair
Started | 272
Completed | 220
Not Completed | 52

BASELINE CHARACTERISTICS:
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 272
Age, Continuous [Median (Full Range); unit: years] | 70 [37 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Secondary and tertiary French care centres
  participants
    France | 272
Body mass index [Median (Full Range); unit: kg/m^2] | 24.8 [16 to 40.4]
Parity [Median (Full Range); unit: children] | 2 [0 to 16]
Post menopause [Count of Participants; unit: Participants] | 257
Hormone replacement therapy [Count of Participants; unit: Participants] | 68
Previous hysterectomy [Count of Participants; unit: Participants] | 58
Previous pelvic organ prolapse surgery [Count of Participants; unit: Participants] | 51
Previous incontinence surgery [Count of Participants; unit: Participants] | 25
Procedure [Count of Participants; unit: Participants]
  Anterior Restorelle® Direct FixTM alone | 95
  Concomitant hysterectomy | 46
  Concomitant posterior Restorelle® Direct FixTM | 63
  Concomitant sub urethral sling | 64
  Concomitant other surgery | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Composite Outcome : Bladder Wound, Rectum Wound, Abnormal Bleeding
Description: Perioperative morbidity
Time Frame: up to 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 272
Participants | 6

2. Secondary Outcome: Number of Patients With Early Complications
Description: Urinary retention, urinary tract infection, hematoma, ureteral complication, second surgery
Time Frame: up to 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 272
Participants | 43

3. Secondary Outcome: Number of Patients With Late Complications
Description: self-catheterization, recurrent urinary tract infections, de novo urinary stress incontinence, chronic pain, vaginal prosthesis exposure, prolapse recurrence, secondary surgery, other
Time Frame: up to 4 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 220
Participants | 43

4. Secondary Outcome: Pelvic Organ Prolapse Quantification (POP-Q) Exam Before Surgery
Description: Pelvic organ prolapse quantification (POP-Q) Staging Criteria Prolapse is staged using POP-Q criteria that can range from good support (no organ descent) reported as a POP-Q stage 0 or I to a POP-Q score of IV (complete procidentia or vault eversion)
Time Frame: preoperative, within 48 hours before surgery
Population: Data was collected retrospectively and few pelvic organ prolapse stage were not available
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 272
Participants
  Cystocele: number analyzed (Participants) | 270
  Cystocele: Stage 0 | 0
  Cystocele: Stage 1 | 1
  Cystocele: Stage 2 | 61
  Cystocele: Stage 3 | 169
  Cystocele: Stage 4 | 39
  Apex: number analyzed (Participants) | 266
  Apex: Stage 0 | 78
  Apex: Stage 1 | 75
  Apex: Stage 2 | 64
  Apex: Stage 3 | 37
  Apex: Stage 4 | 12
  Rectocele: number analyzed (Participants) | 271
  Rectocele: Stage 0 | 115
  Rectocele: Stage 1 | 86
  Rectocele: Stage 2 | 61
  Rectocele: Stage 3 | 5
  Rectocele: Stage 4 | 4

5. Secondary Outcome: Pelvic Organ Prolapse Quantification (POP-Q) Exam After Surgery
Description: as for outcome 4
Time Frame: up to 4 years after surgery
Population: Data was collected retrospectively and few pelvic organ prolapse stage were not available
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 220
Participants
  Cystocele: number analyzed (Participants) | 207
  Cystocele: Stage 0 | 128
  Cystocele: Stage 1 | 54
  Cystocele: Stage 2 | 24
  Cystocele: Stage 3 | 0
  Cystocele: Stage 4 | 1
  Apex: number analyzed (Participants) | 202
  Apex: Stage 0 | 188
  Apex: Stage 1 | 6
  Apex: Stage 2 | 7
  Apex: Stage 3 | 0
  Apex: Stage 4 | 1
  Rectocele: number analyzed (Participants) | 200
  Rectocele: Stage 0 | 174
  Rectocele: Stage 1 | 14
  Rectocele: Stage 2 | 10
  Rectocele: Stage 3 | 2
  Rectocele: Stage 4 | 0

6. Secondary Outcome: Number of Patients With Preoperative Urinary Signs
Description: urinary stress incontinence, overactive bladder, dysuria, masked urinary incontinence
Time Frame: within 4 weeks before surgery
Population: Data was collected retrospectively and few bladder symptom descriptions were not available
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 272
Participants
  Stress urinary incontinence: number analyzed (Participants) | 271
  Stress urinary incontinence | 97
  Overactive bladder: number analyzed (Participants) | 268
  Overactive bladder | 103
  Voiding dysfunction: number analyzed (Participants) | 267
  Voiding dysfunction | 118
  Occult urinary incontinence: number analyzed (Participants) | 259
  Occult urinary incontinence | 48

7. Secondary Outcome: Number of Patients With Postoperative Urinary Signs
Description: urinary stress incontinence, overactive bladder, dysuria, masked urinary incontinence
Time Frame: up to 4 years after surgery
Population: Data was collected retrospectively and few bladder symptom descriptions were not available
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 220
Participants
  Stress urinary incontinence: number analyzed (Participants) | 212
  Stress urinary incontinence | 48
  Overactive bladder: number analyzed (Participants) | 211
  Overactive bladder | 24
  Voiding dysfunction: number analyzed (Participants) | 210
  Voiding dysfunction | 13

8. Secondary Outcome: Number of Patients With Preoperative Digestive Signs
Description: dyschezia, incontinence
Time Frame: within 4 weeks before surgery
Population: Data was collected retrospectively and few bowel symptom descriptions were not available
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 272
Participants
  Dyschezia: number analyzed (Participants) | 256
  Dyschezia | 21
  Faecal incontinence: number analyzed (Participants) | 260
  Faecal incontinence | 13

9. Secondary Outcome: Number of Patients With Postoperative Digestive Signs
Description: dyschezia, incontinence
Time Frame: up to 4 years after surgery
Population: Data was collected retrospectively and few bowel symptom descriptions were not available
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 220
Participants
  Dyschezia: number analyzed (Participants) | 194
  Dyschezia | 6
  Faecal incontinence: number analyzed (Participants) | 188
  Faecal incontinence | 3

10. Secondary Outcome: Number of Patients With Preoperative Active Sexuality
Description: Patients reporting active sexuality
Time Frame: within 4 weeks before surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 198
Participants | 94

11. Secondary Outcome: Number of Patients With Preoperative Dyspareunia
Description: Patients reporting pain
Time Frame: within 4 weeks before surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 87
Participants | 16

12. Secondary Outcome: Number of Patients With Postoperative Active Sexuality
Description: Patients reporting active sexuality
Time Frame: up to 4 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 122
Participants | 41

13. Secondary Outcome: Number of Patients With Postoperative Dyspareunia
Description: Patients reporting pain
Time Frame: up to 4 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 40
Participants | 3

14. Secondary Outcome: Preoperative Score at Numeric Pain Rating Scale
Description: The numeric pain rating scale ranges from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: Within 48 hours before surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 65
units on a scale | 7.3 (1.9)

15. Secondary Outcome: Postoperative Score at Numeric Pain Rating Scale
Description: The numeric pain rating scale ranges from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: up to 48 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Organ Prolapse Repair
Number analyzed (Participants) | 162
units on a scale | 0.46 (0.56)

ADVERSE EVENTS:
Time Frame: The median follow-up was 3 months ranging from 1 to 36 months
Arm/Group | Pelvic Organ Prolapse Repair
All-Cause Mortality (participants affected / at risk) | 0/272
Serious Adverse Events (participants affected / at risk) | 14/272
Other Adverse Events (participants affected / at risk) | 136/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pelvic Organ Prolapse Repair (N=272)
Ureteral injury (Renal and urinary disorders) | 2 — perioperative complication
Urinary tract infection (Renal and urinary disorders) | 2 — perioperative complication
Postoperative haematoma (Renal and urinary disorders) | 2 — postoperative complication in the month following the surgery
3rd degree vaginal prolapse (Renal and urinary disorders) | 7/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
Adverse local tissue reaction around prosthesis (Renal and urinary disorders) | 2/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pelvic Organ Prolapse Repair (N=272)
Bladder injury (Renal and urinary disorders) | 3
Rectal injury (Renal and urinary disorders) | 1
Urinary retention postoperative (Renal and urinary disorders) | 19
Pain (Renal and urinary disorders) | 103
Urinary tract infection (Renal and urinary disorders) | 15
Postoperative haematoma (Renal and urinary disorders) | 6
Chronic pain (Renal and urinary disorders) | 7/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
Adverse local tissue reaction around prosthesis (Renal and urinary disorders) | 8/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
Medical device site granuloma (Renal and urinary disorders) | 6/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
Incontinence (Renal and urinary disorders) | 10/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
1st degree vaginal prolapse (Renal and urinary disorders) | 4/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.
Dyspareunia (Renal and urinary disorders) | 1/220 — Of the 272 patients included, 220 were reviewed at more than one month postoperatively. The description of adverse events is therefore only available for these patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03098641/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03098641/ICF_001.pdf